CLINICAL TRIAL: NCT03549039
Title: Effect of Alveolar Bone Grafting on Health Quality in Patients With Cleft Lip and Palate
Brief Title: Effect of Alveolar Bone Grafting
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Kevser Sancak, research assistant, Ankara University
Other Study IDs: 36290600/22
Record Dates: First submitted 2018-04-08; First posted 2018-06-07 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Alveolar Bone Grafting; Quality of Life
Keywords: quality of life; cleft lip; cleft palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study included patients who underwent secondary alveolar bone grafting by harvesting graft from the anterior iliac crest, in Oral and Maxillofacial Department, Faculty of Dentistry, Ankara University, Turkey, during the period from January 2012 to March 2016. All patients were operated using the same technique and by the same surgical team. Patients will be interviewed to fill Short-Form Health Survey (SF-12) and Postsurgical Patient Satisfaction Questionnaire (PSPSQ) 6 months postoperatively. The questionnaires will be used to assess the relationship between health quality and patient satisfaction. Also, grafted sites will be evaluated with respect to fistula, the presence of cleft palate, and infection.The descriptive statistics and Pearson correlation analyses will be made using PSPSQ scores and SF-12 PCS and MCS scores.

DETAILED DESCRIPTION:
The postsurgical patient satisfaction questionnaire (PSPSQ) was designed to assess each patient's overall satisfaction with the procedure(s), functional improvements, and recognized or perceived negative effects of the procedures. One of the most commonly used measures of HRQoL is SF-36, which has been reduced to 12 items with the minimal loss of information to form SF-12 . HRQoL was assessed using SF-12 Physical Component Summary (PCS) and Mental Component Summary (MCS) scores.

ELIGIBILITY:
Inclusion Criteria:

patients who were undergone alveolar cleft surgery before at our hospital at least 6 months after surgery

Exclusion Criteria:

patients who don't accept to join questionnaire

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent surgery due to alveolar cleft
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Short-Form Health Survey (SF-12) Physical Component Summary | 20 minutes
  all participants will be called to faculty. SF-12 will be done. SF-12 is calculated using the scoring table. Health-related quality of life, which was measured using the Physical Component Summary (PCS) scores of SF-12 was assessed. Physical component is scored from 0 to 100 with 0 representing the worst and 100 representing the best health status.
Short-Form Health Survey (SF-12) Mental Component Summary | 20 minutes
  all participants will be called to faculty. SF-12 will be done. SF-12 is calculated using the scoring table. Health-related quality of life, which was measured using the Mental Component Summary (MCS)scores of SF-12 was assessed. Mental component is scored from 0 to 100 with 0 representing the worst and 100 representing the best health status.
Postsurgical Patient Satisfaction Questionnaire (PSPSQ) | 20 minutes
  all participants will be called to faculty. PSPSQ will be done. Patient satisfaction will be assessed by analyzing data gathered from PSPSQ. PSPSQ included seven questions. It is designed to assess each patient's overall satisfaction with the procedure(s), functional improvements, and recognized or perceived negative effects of the procedures. The 7-point Likert (poor to excellent), scale is used so that the person who answers the questions can rate the level of related satisfaction with each question. The final outcome is between 7 and 49. Higher scores are associated with satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Sancak, Study Chair — Ankara University Faculty of Dentısry
Locations (1):
- Ankara University dentisry of faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
de-identified individual participant data for all primary and secondary outcome measures will be made available

REFERENCES:
- [Background] Rustemeyer J, Gregersen J. Quality of Life in orthognathic surgery patients: post-surgical improvements in aesthetics and self-confidence. J Craniomaxillofac Surg. 2012 Jul;40(5):400-4. doi: 10.1016/j.jcms.2011.07.009. Epub 2011 Aug 23. PMID 21865051
- [Background] Gandhi SK, Salmon JW, Zhao SZ, Lambert BL, Gore PR, Conrad K. Psychometric evaluation of the 12-item short-form health survey (SF-12) in osteoarthritis and rheumatoid arthritis clinical trials. Clin Ther. 2001 Jul;23(7):1080-98. doi: 10.1016/s0149-2918(01)80093-x. PMID 11519772
- [Background] Motegi E, Hatch JP, Rugh JD, Yamaguchi H. Health-related quality of life and psychosocial function 5 years after orthognathic surgery. Am J Orthod Dentofacial Orthop. 2003 Aug;124(2):138-43. doi: 10.1016/s0889-5406(03)00391-3. PMID 12923507